CLINICAL TRIAL: NCT05057247
Title: A Phase II Study of Duvelisib Plus Docetaxel in PD-1 Inhibitor Experienced Patients With Incurable Head and Neck Squamous Cell Carcinoma
Brief Title: Duvelisib Plus Docetaxel In Recurrent/Metastatic HNSCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glenn J. Hanna (Other)
Collaborators: Secura Bio, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Glenn J. Hanna, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-393
Record Dates: First submitted 2021-09-08; First posted 2021-09-27 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck (SCCHN); Recurrent Squamous Cell Carcinoma of the Head and Neck; Metastatic Head and Neck Cancer; Advanced Head and Neck Cancer; Advanced Head and Neck Squamous Cell Carcinoma
Keywords: Squamous cell carcinoma of the head and neck (SCCHN); Recurrent Squamous Cell Carcinoma of the Head and Neck; Metastatic Head and Neck Cancer; Advanced Head and Neck Cancer; Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — duvelisib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Duvelisib plus Docetaxel chemotherapy (Experimental): Participants will receive duvelisib by mouth twice daily,dosage per protocol continuously (days 1-21 of a 21-day cycle) with a 7-day lead-in planned prior to the start of taxane therapy.
  Docetaxel at via IV will be delivered on day 1 of each 21-day cycle.
  Treatment will continue for 24-months or until unacceptable toxicity, progression, or death.
  Interventions: Drug: Duvelisib; Drug: Docetaxel

INTERVENTIONS:
Drug: Duvelisib — Duvelisib capsules should be swallowed whole with a glass of water (approximately 8 ounces).
  Advise patients not to open, break, or chew the capsules. Duvelisib may be administered without regard to meals; however, subjects should avoid grapefruit and grapefruit juice while on duvelisib.
  continue for up to 24 months.
  Other Names: VS-0145
Drug: Docetaxel — Docetaxel chemotherapy once every 21 days (by intravenous infusion) over about 30- 60 minutes at each visit. This will continue for up to 24 months
  Other Names: Taxotere

SUMMARY:
This trial that is investigating a medication called duvelisib in combination with docetaxel for the treatment of squamous cell carcinoma of the head and neck (SCCHN) that has returned or spread outside the head and neck area.

The names of the study drugs involved in this study are:

* Duvelisib (PI3K inhibitor)
* Docetaxel chemotherapy

DETAILED DESCRIPTION:
This multicenter, phase II open-label, single-arm trial will enroll participants with recurrent or metastatic (R/M), incurable squamous cell carcinoma of the head and neck (SCCHN) who have failed or discontinued PD-1 blockade in the first-line (1L) advanced disease setting, regardless of human papillomavirus (HPV) and smoking status, or PI3K pathway alteration status.

This research study involves the oral (taken by mouth) agent duvelisib with the intravenous (IV) chemotherapy agent docetaxel.

The names of the study drugs involved in this study are:

* Duvelisib (PI3K inhibitor)
* Docetaxel chemotherapy

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will receive study treatment for up to 2 years and will be followed for 3 years.

It is expected that about 30 people will take part in this research.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug (duvelisib) to learn whether it works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved duvelisib for this specific disease but has approved it for other uses (such as certain types of blood cancers). The FDA has approved docetaxel as a treatment option for head and neck cancer, as well as other cancer types.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Participants must have histologically confirmed squamous cell carcinoma of the head and neck (SCCHN) with evidence of recurrent, metastatic (R/M) or advanced, incurable disease from any mucosal subsite including oral cavity, oropharynx, larynx, hypopharynx, nasal cavity, and the paranasal sinuses.
* Participants must have at least one RECIST v1.1 measurable lesion, as defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) ≥1 cm with CT scans or MR imaging.
* Must have had at least 1, but no more than 2, prior lines of prior systemic therapy for R/M SCCHN; one of these lines should have included PD-1/L1 blockade

  * Platinum-based therapy as part of definitive/adjuvant or curative-intent treatment can count as 1 prior line of therapy if the subject progressed within 6 months of receiving therapy.
  * At least 2 weeks must have elapsed since the end of prior chemotherapy, biological agents (3 weeks for anti-cancer monoclonal antibody containing regimens) or any investigational drug product, with adequate recovery of treatment-related toxicity to NCI CTCAE Version 5.0 grade ≤1 (or tolerable grade 2) or back to baseline (except for alopecia or peripheral neuropathy).
* Be ≥18 years of age on the day of signing informed consent.
* Must provide prior data on tumor PD-L1 expression status and HPV status, if available
* Have a performance status of 0 or 1 on the ECOG Performance Scale
* Participants must have adequate organ and marrow function as defined below (within 14 days prior to study registration):

  * absolute neutrophil count ≥ 1,000/mcL
  * hemoglobin ≥ 9 g/dL
  * platelets ≥ 100,000/mcL
  * total bilirubin ≤ upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5x institutional ULN (or ≤ 1.5x institutional ULN if concomitant with alkaline phosphatase >2.5x institutional ULN) or ≤ 5x ULN for those with liver metastases
  * serum creatinine ≤ 1.5x ULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above 1.5x ULN
  * coagulation profile INR ≤ 1.5x ULN unless the participant is receiving an anticoagulant
* Baseline tumor measurements must be documented from imaging within 28 days prior to study registration.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 7 days of study registration. Female subjects of childbearing potential should have a negative urine or serum pregnancy test repeated within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female and male subjects of childbearing potential must agree to use an adequate method of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 4 months after completion of stud drug administration. Contraception is required before starting the first dose of study medication through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Be willing and able to provide written informed consent for the trial.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Have been previously treated with 3 or more lines of systemic therapy for R/M SCCHN.

  -- Have received treatment with a prior PI3K pathway inhibitor
* Have received radiation therapy (RT) within 14 days of the first dose of duvelisib on study.
* Participant has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging and off systemic steroids for at least 4 weeks prior to the first dose of study treatment), and have no evidence of new or enlarging brain metastases. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability, because of the poor prognosis and progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Concurrent administration of other cancer specific therapy or investigational agents during the course of this study.
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection; evidence of symptomatic congestive heart failure, unstable angina pectoris, stroke, or ventricular arrhythmia within 6 months of enrollment.
* Have received a live or live attenuated vaccine within 4 weeks of the first dose of duvelisib.
* Have received medications or consumed foods that are strong inhibitors or inducers of cytochrome P450 (CYP3A) within 2 weeks of, or while on, duvelisib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J. Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from Octorber 14, 2021 to October 10, 2023.
Groups:
- Duvelisib Plus Docetaxel Chemotherapy: Patients received duvelisib at the same dose of 25mg orally twice daily on days 1 through 21. Docetaxel was administered intravenously (IV) at a dose of 75 mg/m2 on day 1 of a 21-day cycle. Treatment duration is planned for 24 months (or longer if patient exhibits good tolerance and clinical benefit), unless unacceptable toxicity, disease progression, or withdrawl of consent occurs. Following the first 21-day cycle of therapy, both duvelisib and docetaxel are to be continued concurrently in 21-day subsequent cycles.
Period: Overall Study
Arm/Group | Duvelisib Plus Docetaxel Chemotherapy
Started | 26
Completed | 0
Not Completed | 26
Not completed — Death | 4
Not completed — Physician Decision | 3
Not completed — Progressive Disease | 7
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 6
Not completed — Subject Non-Compliance | 1
Not completed — On treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Duvelisib Plus Docetaxel Chemotherapy
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (64.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 11
    1 | 15
PD-L1 Status (pre-treatment) [Count of Participants; unit: Participants]
  Negative (CPS 0 to <1) | 2
  Positive (CPS 1 or greater) | 22
  Unknown | 2
TP53 status (pre-treatment) [Count of Participants; unit: Participants]
  Mutated | 10
  Negative | 16
PI3K statue (Pre-treatment） [Count of Participants; unit: Participants]
  Negative | 19
  Positive | 7
Primary Disease Site at Initial Diagnosis [Count of Participants; unit: Participants]
  Hypopharynx | 2
  Larynx | 1
  Oral Cavity | 11
  Oropharynx | 12
Site of recurrence prior to registration [Count of Participants; unit: Participants]
  Locoregional | 6
  Distant | 10
  Both | 10
HPV status [Count of Participants; unit: Participants]
  Negative | 12
  Positive | 14
Smoking History [Count of Participants; unit: Participants]
  No | 8
  Yes | 18
Current Smoker [Count of Participants; unit: Participants]
  No | 18
  Yes | 3
  Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR) Rate
Description: BOR rate was defined as the proportion of participants that experienced complete response (CR) or partial response (PR) on treatment based on RECIST 1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Median time on treatment was 2.3 months (range 0.7-21.9 months)
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Duvelisib Plus Docetaxel Chemotherapy
Number analyzed (Participants) | 26
proportion of participants | 0.19 [0.068 to 0.41]

2. Secondary Outcome: Median Overall Survival (OS)
Description: OS based on the Kaplan-Meier method was defined as the time from registration to death due to any cause, or censored at date last known alive.
Time Frame: The median follow-up time was 6.5 months (range 0.7 - 26 months).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Duvelisib Plus Docetaxel Chemotherapy
Number analyzed (Participants) | 26
Months | 10.2 [6.7 to 15.9]

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS based on the Kaplan-Meier method was defined as the time from registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: Median follow-up time was 2.3 months (range 0.7-21.9 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Duvelisib Plus Docetaxel Chemotherapy
Number analyzed (Participants) | 26
Months | 2.8 [1.9 to 7.0]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Median follow-up time was 2.3 months (range 0.7-21.9 months)
Population: Only participants who have responded to the treatment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Duvelisib Plus Docetaxel Chemotherapy
Number analyzed (Participants) | 5
Months | 5.1 [0.7 to 15.5]

5. Secondary Outcome: Number of Participants With Treatment Related Adverse Events Per CTCAE 5.0
Description: The number of participants who experienced the treatment-related adverse events per CTCAE 5.0 during the time of treatment.
Time Frame: Median follow-up time was 2.3 months (range 0.7-21.9 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib Plus Docetaxel Chemotherapy
Number analyzed (Participants) | 26
Participants | 25

6. Secondary Outcome: Change of QLQ H&N 35 From Cycle 1 to Cycle 4
Description: The QLQ H&N35 incorporates seven multi-item scales that assess pain, swallowing, senses (taste and smell), speech, social eating, social contact and sexuality. There are also eleven single items. The score range from 0 to 100.
  For all items and scales, high scores indicate more problems, so negative difference indicates better QoL (less problems) at C4D1 compared to C1D1.
Time Frame: Up to 3 months
Population: The analysis population included the patients who answered at least some questions at both cycle 1 day 1 and cycle 4 day 1.
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Duvelisib Plus Docetaxel Chemotherapy
Number analyzed (Participants) | 11
Units on a scale
  Pain | -3.8 [-25 to 16.7]
  Swallowing | -1 [-25 to 30.6]
  Senses problems | 7.6 [-16.7 to 50]
  Speech problems | 4.5 [-11.1 to 50]
  Trouble with social eating | 0.76 [-16.7 to 16.7]
  Trouble with social contact | -1.2 [-20 to 13.3]
  Less sexuality | 6.1 [0 to 33.3]
  Teeth | -6.1 [-33.3 to 0]
  Opening mouth | 9.1 [-33.3 to 33.3]
  Dry mouth | 60.6 [0 to 100]
  Sticky saliva | -6.7 [-33.3 to 0]
  Coughing | 9.1 [-33.3 to 33.3]
  Felt ill | 0 [-33.3 to 33.3]

ADVERSE EVENTS:
Time Frame: Median follow-up time for adverse events was 2.3 months (range 0.7-21.9 months). Median follow-up time for survival was 6.5 months (range 0.7 - 26 months).
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose, results in death; is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is an important medical event,suspected transmission of an infectious agent via the study drug is an SAE.
Arm/Group | Duvelisib Plus Docetaxel Chemotherapy
All-Cause Mortality (participants affected / at risk) | 17/26
Serious Adverse Events (participants affected / at risk) | 10/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib Plus Docetaxel Chemotherapy (N=26)
Cardiac arrest (Cardiac disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Edema face (General disorders) | 1
Fever (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Thrush (Infections and infestations) | 1
Viremia (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Weight loss (Investigations) | 1
Hyperlipidemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib Plus Docetaxel Chemotherapy (N=26)
Anemia (Blood and lymphatic system disorders) | 26
Lymph node pain (Blood and lymphatic system disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Conduction disorder (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 7
Tinnitus (Ear and labyrinth disorders) | 5
Endocrine disorders - Other, specify (Endocrine disorders) | 6
Hypothyroidism (Endocrine disorders) | 17
Testosterone deficiency (Endocrine disorders) | 1
Dry eye (Eye disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 1
Periorbital edema (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 12
Dental caries (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 15
Dry mouth (Gastrointestinal disorders) | 15
Dyspepsia (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 15
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 14
Oral pain (Gastrointestinal disorders) | 5
Rectal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Disease progression (General disorders) | 1
Edema face (General disorders) | 3
Edema limbs (General disorders) | 7
Facial pain (General disorders) | 2
Fatigue (General disorders) | 23
Fever (General disorders) | 2
Gait disturbance (General disorders) | 2
General disorders and administration site conditions - Other, specify (General disorders) | 1
Localized edema (General disorders) | 1
Malaise (General disorders) | 1
Neck edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 2
Autoimmune disorder (Immune system disorders) | 1
Hepatic infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Salivary gland infection (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Thrush (Infections and infestations) | 3
Tooth infection (Infections and infestations) | 1
Viremia (Infections and infestations) | 3
Bruising (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 4
Fracture (Injury, poisoning and procedural complications) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 24
Alkaline phosphatase increased (Investigations) | 15
Aspartate aminotransferase increased (Investigations) | 23
Blood bilirubin increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Creatinine increased (Investigations) | 16
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
INR increased (Investigations) | 1
Lipase increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 8
Serum amylase increased (Investigations) | 1
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hyperlipidemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 5
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysarthria (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Memory impairment (Nervous system disorders) | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 8
Somnolence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 3
Irritability (Psychiatric disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 2
Erectile dysfunction (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 2
Nail changes (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 24
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 11
Hypotension (Vascular disorders) | 2
Lymphedema (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT05057247/Prot_SAP_000.pdf